CLINICAL TRIAL: NCT00496275
Title: A Phase I, Open Label Study to Assess the Safety and Tolerability of ZD6474 (ZACTIMA) in Combination With Vinorelbine (Navelbine) or Gemcitabine (Gemzar) Plus Cisplatin as First Line Therapy in Patients With Locally Advanced or Metastatic (Stage IIIB-IV) Non Small Cell Lung Cancer.
Brief Title: Phase I Combination With Vinorelbine or Gemcitabine Plus Cisplatin in Locally Advanced or Metastatic NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00054
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; ZACTIMA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Vinorelbine; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zactima (ZD6474)
Drug: Vinorelbine plus cisplatin
Drug: Gemcitabine plus cisplatin

SUMMARY:
To test the safety and tolerability of ZD6474 in combination withVinorelbine (Navelbine) or Gemcitabine (Gemzar) plus cisplatin as first line therapy in patients with locally advanced or metastatic (Stage IIIB-IV) Non Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed non small cell lung cancer (stage IIIB-IV)
* Life expectancy greater than 12 weeks
* At least 1 measurable lesion greater than 10mm in smallest diameter.

Exclusion Criteria:

* Prior treatment with anticancer agent
* Brain metastases
* Major surgery within last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Establish safety and tolerability of ZACTIMA in combination with vinorelbine plus cisplatin or gemcitabine plus cisplatin

SECONDARY OUTCOMES:
Pharmacokinetics of ZACTIMA, vinorelbine or gemcitabine, plus cisplatin when co-administered | Predetermined timepoints after dose administration
Preliminary assessment of efficacy of ZACTIMA when co-administered with vinorelbine plus cisplatin or gemcitabine plus cisplatin

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi